CLINICAL TRIAL: NCT07283978
Title: Real-world Exploration of Digital iNnovation in the Management of Excess Weight
Acronym: RENEW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 351778
Record Dates: First submitted 2025-11-19; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Obesity
Keywords: Weight Management; Digital Weight Management; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: All participants will receive the same intervention but at different times during their obesity treatment. Group A will receive the intervention while waiting to start standard of care weight management services and Group B will receive the intervention upon discharge from their standard of care weight management services.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A Intervention (Active Comparator): Study participants who receive 12 months of digital weight management services delivered through a smartphone app.
  Interventions: Other: Digital Weight Management Programme
- Group B Intervention (Active Comparator): Study participants who receive 12 months of digital weight management services delivered through a smartphone app
  Interventions: Other: Digital Weight Management Programme
- Group A Controls (No Intervention): Patients who receive standard of care weight management services
- Group B Controls (No Intervention): Patients who receive standard of care service after discharge from standard of care weight management services

INTERVENTIONS:
Other: Digital Weight Management Programme — Digital Weight Management Programme
  Arms: Group A Intervention; Group B Intervention

SUMMARY:
This is a real-world study. The purpose of this research is to explore whether a new National Institute for Health and Care Excellence (NICE)-approved digital weight-management model of care can improve health service delivery and address the Quintuple Aim of Healthcare (health outcomes, cost, patient and clinician experience, and health inequalities), for individuals living with obesity accessing National Health Service (NHS) Tier 3 weight-management services.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Referred to South east London Tier 3 weight management pathway by their GP
* Accepted by the GSTT Tier 3 weight management service

Exclusion Criteria:

* Participants is Group A cannot participate in Group B
* Do not have use of a smartphone
* Do not read, write, or speak English
* Are unable and/or unwilling to provide informed consent
* Have a diagnosis of an eating disorder
* Have had bariatric surgery
* Currently have deranged thyroid function tests (required as part of normal referral process)
* Have type-1 diabetes
* Are on insulin or sulfonylureas at high risk of hypoglycaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of weight change at 12 months | Baseline and 12 months
Quality of Life as a measure to determine cost-effectiveness | Baseline and 12 months
  Quality of Life will be measured using the European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) questionnaire

SECONDARY OUTCOMES:
Feasibility of implementing the intervention into Tier 3 weight management pathways | Once
  This will be assessed through qualitative interviews with participants in the Sub-study.
Acceptability of implementing the intervention into Tier 3 weight management pathways | Once
  This will be assessed through qualitative interviews with participants in the Sub-study.
Uptake of the intervention | 12 months
Retention in the intervention programme | From enrolment until the end of the intervention at 12 months /withdrawal/dropout
Success in the intervention programme | From enrolment until the end of the intervention at 12 months
  This will be assessed as clinically significant percentage in weight change of greater than or equal to 5 percent.
Economic measurements - Quality of Life Years | Baseline, 6 months, and 12 months
  Quality-Adjusted Life Years (QALYs) associated with weight loss, calculated from the scores on the European Quality of Life 5 Dimensions Level questionnaire (EQ-5D-5L)
Economics measurements - Resource Use | From enrolment to the end of the intervention at 12 months
  Resource use covering primary and secondary care services within the National Health Service (NHS)
Economics measurements - Unit costs | From enrolment to end of intervention at 12 months
  Unit costs obtained from standard sources such as NHS reference costs and Personal Social Services Research Unit's unit costs for health and social care.
Economics measurements - Costs between intervention group and standard care group | From enrolment to end of intervention at 12 months
  Costs between intervention group and standard care group with be compared
Patient reported outcomes - alcohol use | At Baseline, 6 months, and 12 months
  This will be assessed using a self-reported questionnaire - Alcohol Use Disorders Identification Test (Audit) / scale ranges 0 - 40 / 0=low risk, 20 or more = possible alcohol dependence
Patient reported outcomes - patient health | Baseline, 6 months, 12 months
  This will be assessed using the self-reported Patient Health Questionnaire-4 (PH-4) / Score range 0 - 12) / Score of 3 or higher further assessment for depression &/or anxiety recommended
Patient reported outcomes - eating pattern | Baseline, 6 months, 12 months
  This will be assessed using the self-reported Three-Factor Eating Questionnaire / Score range 1 - 4 for each question / scores are summated into scale scores for cognitive restraint, uncontrolled eating, and emotional eating.
Patient reported outcomes - binge eating | Baseline
  This will be assessed using the self-reported Binge Eating Scale (BES) questionnaire / Score range 0 - 46 / 17 or lower = low binge-eating, 18-26 = mild to moderate binge-eating, 27 or higher = severe binge-eating
Patient reported outcomes - physical activity | Baseline if required per clinician assessment
  This will be assess using the self-reported General Practice Physical Activity Questionnaires / Scoring is: Inactive, Moderately inactive, Moderately active, or Active
Sub-group analyses- Use of glucagon-like peptide (GLP-1) agonists | From enrolment until the end of intervention at 12 months
  Participant use (never/commenced during study/used throughout) of GLP-1 agonsits will be assessed
Sub-group analyses - Adherence | From enrolment until drop-out, withdrawal, or end of intervention at 12 months
  Participant adherence to the intervention will be assessed
Sub-group analyses - Comorbidities | From enrolment until end of intervention at 12 months
  Obesity-related medical comorbidities will be assessed
Sub-group analyses - Social demographics | At enrolment
  Participant social demographics such as sex, ethnicity, age, and Index of Multiple Deprivation (IMD) will be assessed.
Clinical measures - height | Baseline
  Height in metres will be assessed as part of the clinical measures analysis
Clinical measures - blood pressure | Baseline, 6 months, and 12 months
  Self-reported blood pressure will be assessed as part of the clinical measures analysis
Clinical measures - Body Mass Index | Baseline, 6 months, and 12 months
  Body Mass Index (BMI) will be assessed from self-reported weight in kilograms divided by height in metres squared, as part of the clinical measures analysis.
Clinical Measures - waist circumference | Baseline, 6 months, 12 months
  Self-reported waist circumference in centimetres will assessed as part of the clinical measures analysis

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Walker, PhD, Study Chair — Guy's and St Thomas NHS Foundation Trust; Emma Duncan, MD, PhD, Study Director — King's College London
Locations (1):
- Guy' & St Thomas' NHS Foundation Trust, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided